CLINICAL TRIAL: NCT06429527
Title: Evaluating App-Based Vision Testing (WHOeyes) Combined with the Questionnaire As a Substitute for One-Week Postoperative In-Clinic Follow-Up in Age-Related Cataract Patients: a Multi-center Randomized Controlled Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Eye & ENT Hospital of Fudan University (Other); Shenzhen Eye Hospital (Other); The Eye Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Beijing Tongren Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Lixia Luo, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024KYPJ037
Record Dates: First submitted 2024-05-09; First posted 2024-05-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-11

CONDITIONS: Cataract Senile
Keywords: cataract; telemedicine; health economics; carbon emission; follow-up postoperatively
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote follow-up (Experimental): One week postoperatively, the participants use the WHOeyes app to test their uncorrected visual acuity and fill in a self-made discomfort identification questionnaire.
  Visit the clinics for review 1 day and 1 month post-cataract surgery.
  Interventions: Behavioral: WHOeyes combined with a questionnaire.
- Usual care (No Intervention): Participants routinely returned to the hospital for review 1 day, 1 week and 1 month post-cataract surgery

INTERVENTIONS:
Behavioral: WHOeyes combined with a questionnaire. — The WHOeyes app (a self-administered visual acuity testing app) plus a questionnaire (to ask the patients to go to the hospital if they ever experience ocular discomfort including eye redness, discharge, etc.) will be used for 1-week follow-up after cataract surgery, and only those with significant vision loss based on WHOeye test or with ocular discomfort are advised to return to the hospital for follow-up.
  Arms: Remote follow-up

SUMMARY:
The goal of this clinical trial is to learn if an app-based vision testing (WHOeyes) combined with a questionnaire can recognize those who have to go back to the hospital, and thus replace the in-clinic 1-week review after an uncomplicated cataract surgery in people with senile cataract. It will also learn about the cost-effectiveness and environmental benefits of such remote follow-up pattern. Besides, the safety and user's satisfaction will also be evaluated. The main questions it aims to answer are:

For people with uncomplicated senile cataract, does 1-week clinical follow-up replaced with remote follow-up (using a vision test app and a questionnaire) not adversely affect patients' prognosis? Can this alternative approach bring greater cost-effectiveness and environmental friendliness compared to the traditional follow-up method? Researchers will compare one-week remote follow-up to a routine clinical follow-up to see if one-week remote follow-up is feasible.

Participants will:

Visit the clinic to finish routine follow-up 1 day and 1 month after cataract surgery.

Using app (WHOeyes) and a questionnaire at home or visit the clinic 1 week after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Senile cataract patients undergoing Phaco + IOL implantation under local anesthesia.
2. Between 50 and 80 years of age, regardless of gender.
3. The subject or their family members own a smartphone, understand and can correctly install and use the WHOeyes app for vision testing under the guidance of a physician.
4. Able to understand and cooperate with the trial procedures, voluntarily participate in this clinical trial, and sign an informed consent form.

Exclusion Criteria:

1. Had other serious eye diseases in addition to cataract, including:

   1. Chronic or recurrent eye diseases of the study eye, such as keratitis or corneal malnutrition, iritis, scleritis, uveitis, iridocyclitis. (Note: refractive errors, dry eye, chronic conjunctivitis, and mild pterygium are not exclusionary.
   2. Active ocular infection or inflammation in either eye.
   3. Episode of acute uveitis within the past 6 months in either eye.
   4. Intraocular pressure >21mmHg or a history of glaucoma in the study eye.
   5. Presence of unstable active lesions or other ocular diseases of the study eye that, in the investigator's judgment, could potentially interfere with the study evaluation or compromise subject safety (e.g., moderate to severe diabetic retinopathy, wet age-related macular degeneration, retinal detachment).
   6. Congenital abnormalities in the study eye (e.g., congenital cataracts, aniridia).
   7. Corrected visual acuity in the non-study eye <0.1 (20/200).
2. History of ocular trauma in the study eye.
3. History of ocular surgery in the study eye, such as glaucoma surgery, vitrectomy, corneal refractive surgery, corneal transplantation.
4. Scheduled ocular surgery in either eye during the study period, such as trabeculectomy, corneal transplantation.
5. Occurrences of intraoperative and postoperative complications (e.g., elevated intraocular pressure, corneal edema) in the study eye within 1 day after cataract surgery.
6. Corrected visual acuity of the study eye less than 0.5 (20/40) on postoperative day 1.
7. With severe chronic systemic diseases or are susceptible to infection, including:

   1. Poorly controlled diabetes (fasting blood glucose >10 mmol/L).
   2. Poorly controlled hypertension (systolic blood pressure>160mmHg or diastolic blood pressure>100mmHg).
   3. Ongoing systemic treatment for infectious diseases;
   4. Presence of cachexia or bone marrow suppression.
   5. Confirmed diagnosis of AIDS or positive test results for HIV antibodies.
   6. Presence of severe cardiovascular, pulmonary, hepatic, renal, endocrine, immune, dermatological, musculoskeletal, neurological, or psychiatric diseases, hearing impairment, or mobility impairment, as deemed unsuitable for participation in this trial by the investigator.
8. Participation in other clinical trials within the last 30 days (excluding those who only participated in screening process without receiving any investigational drugs or devices).
9. Have pre-planned hospital visits during the study period, other than those required for postoperative follow-ups of the study eye;
10. Any other condition or circumstance that, in the investigator's judgment, makes the patient unsuitable for participation in this trial.

Note: The study eye refers to the eye that underwent cataract surgery and is included in this study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The best corrected distant visual acuity (BCVA) of the operative eye | 1 month after cataract surgery
  Using the ETDRS chart to test the BCVA of the operative eye.

SECONDARY OUTCOMES:
Incremental cost-effectiveness ratios (ICERs) | 1 month postoperatively
  Mean difference in costs divided by mean difference in quality adjusted life years (QALYs).
Carbon emission | 1 week and 1 month postoperatively
  Collect the carbon emission related activity data generated in the process of postoperative follow-up of patients and hospital through enquiry and questionnaire.
Uncorrected distant visual acuity (UDVA)of the operative eye | 1 month postoperatively
  Using the ETDRS chart to test the UDVA of the operative eye.
Incidence and severity of postoperative complications | Until 1 month postoperatively
  The proportion of postoperative complications of cataract in the two groups 1 week after surgery was calculated, and the postoperative complications were diagnosed by professional doctors.
Incidence and severity of self-reported ocular discomfort | Until 1 month postoperatively
  Collected by self-reported outcomes and past medical records (if any) of subjects.
Number of unplanned visits | Until 1 month after cataract surgery
  Collected by self-reported outcomes and past medical records (if any) of subjects.
Patient reported outcome measures (PROMs): Catquest-9SF | 1 month after cataract surgery
  Vision-specific quality of life is measured by the Chinese version of 9-item short-form of Catquest questionnaire (Catquest-9SF). There are five text response options for the answers scaled from "Yes, very great difficulties" to "No, no difficulties" including answer "Cannot decide". The minimum score is 9 and maximum score is 36, and lower scores mean a better outcome.
Patient reported outcome measures (PROMs): NEI-VFQ-25 | 1 month after cataract surgery
  Vision-specific quality of life as measured by the Chinese version of National Eye Institute Visual Function Questionnaire (NEI-VFQ-25). The minimum score is 0 and maximum score is 100, and higher scores mean a better outcome.
Patient reported outcome measures (PROMs): EQ-5D-5L | 1 month after cataract surgery
  Health-related quality of life as measured by the Chinese version of five-level EuroQol five-dimensional questionnaire (EQ-5D-5L). The overall answer for the five dimensions can be combined into a five-digit number that describes the patient's health state. The raw scores are also converted to an EQ-5D index value (Chinese value set) ranging from -0.391 (worst perceived health state) to 1 (best perceived health state).
Users' satisfaction with the WHOeyes app | 1 month after cataract surgery
  Assessed by a self-made questionnaire, the answer of it can converted into a 5-point scale. The minimum value is 1 and the maximum value is 5. The higher the scores are, the greater the satisfaction the users have.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No